CLINICAL TRIAL: NCT05368142
Title: The Clinical Efficacy and Safety of Topical Nocardia Cell Wall Skeleton in the Treatment of Diabetic Foot Ulcer Wounds- A Prospective, Randomized, Controlled, Multicentre Study
Brief Title: Nocardia Cell Wall Skeleton for the Treatment of Diabetic Foot Ulcer Wounds
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: Gulou Hospital Affiliated to Medical College of Nanjing University (Unknown); Suzhou Municipal Hospital (Other); Affiliated Hospital of Nantong University (Other); Affiliated Hospital of Jiangnan University (Other); Huai'an First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XYFY2021-KL151-01
Record Dates: First submitted 2021-07-27; First posted 2022-05-10 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-01

CONDITIONS: Diabetic Foot Ulcer; Therapy, Directly Observed
Keywords: Diabetic Foot Ulcer; Nocardia Rubra Cell Wall Skeleton
MeSH Terms: conditions — Diabetic Foot; Directly Observed Therapy | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-CWS treatment group (Experimental): Patients with N-CWS treatment
  Interventions: Drug: Nocardia rubra Cell Wall Skeleton
- Control group（ treatment with Silver Ion-releasin) (Placebo Comparator): Patients with Silver Ion-releasin
  Interventions: Drug: Silver ions dressing

INTERVENTIONS:
Drug: Nocardia rubra Cell Wall Skeleton — Nocardia rubra cell wall skeleton for external application
  Other Names: Treatment group
  Arms: N-CWS treatment group
Drug: Silver ions dressing — Silver ions dressing for external application
  Other Names: Control group
  Arms: Control group（ treatment with Silver Ion-releasin)

SUMMARY:
This study was to investigate the efficacy and safety of Nocardia rubra Cell Wall Skeleton (NCWS) in the treatment of diabetic foot ulcer wounds. The study was a prospective, randomized, controlled, multicentre study . The subjects were randomly divided into two groups: NCWS group and control group（silver ions dressing）, with a total of 116 cases and 58 cases in each group. Patients in the NCWS group received nocardia rubra cell wall skeleton for external use, in parallel with silver ions dressing treatment. The efficacy and side effects were observed, with a primary endpoint of 30-days wound healing rate.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 to 80 years old (including 18 and 80 years of age), gender not limited;
* in patients with type 2 diabetic foot, in 1999 the WHO diagnostic criteria, diabetic foot screening period or three months before randomization glycated hemoglobin (HbA1C) was detected in 10% or less;
* the target body ankle brachial index of at least 0.8, without intermittent claudication walkers;
* the target ulcer must have the following characteristics: A) according to the Wagner ulcer classification system for level 1 or level 2 B) ulcer is located in the foot, ankle and shin before; C) wound area of 2-5 cm2; D) has existed at least 4 weeks before randomization; E) if you have multiple wounds, select into the set standard and area is one of the biggest intervention and evaluation of the wound.The rest of the wound conventional treatment is not included in the study;If there are two or more wounds are the biggest, choose the worst into classification research;If there are two or more wound area and the classification, choice wound area are the longest study; F) without visible pus and necrotic material;
* voluntary to participate in this clinical study, cooperate a doctor to conduct research, and sign the informed consent.

Exclusion Criteria:

* with clear surgical indications, such as vascular occlusion, bone exposed, abscess, osteomyelitis, etc;
* into the group of the first 3 months of vascular reconstruction or angioplasty;
* impaired liver function (ALT and AST 3 times more than normal limit, AST, aspartate amino transferase;ALT: alanine aminotransferase);
* serum creatinine greater than 2 times the upper limit of normal value;
* serum albumin < 2.0 g/dL;
* is undergoing immunosuppressive medication;
* Various malignant tumor patients ;
* of pregnant women, nursing mothers, or in the near future with family planning; ● with nerve, mental disorders and can't cooperation or unwilling to partners, has a history of alcoholism, drug abuse, and failed to quit;
* into the group of the first 3 months participated in other clinical subjects; Cartesian bacteria cell wall
* to use red, skeleton or silver products are taboo, allergies or known allergies;
* researchers believe that patients should not participate in this study to other situations.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-05-20 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Wound healing rate up to 30 days | 30 days after first medicine application
  The wound healing rate for 30 days treatment（physiological parameter）

SECONDARY OUTCOMES:
Healing time | From date medicine application until the complete closure of wound, assessed up to 30 days
  The time with complete closure of wound within 30 days treatment
Healing rate | 30 days after first medicine application
  The rate of complete closure of wound for 30 days treatment
Surgical intervention rate | From first medicine application to 30 days
  The rate of Surgical intervention for 30 days treatment（physiological parameter）
Pathogenic bacteria positive rate | 30 days after first medicine application
  The rate of Pathogenic bacteria positive for 30 days treatment（physiological parameter）

IPD SHARING:
Plan to Share IPD: No